CLINICAL TRIAL: NCT00196157
Title: Linear Anatomically Versus Focal Electrophysiologically Guided Substrate Ablation in Patients With Persistent Atrial Fibrillation
Brief Title: Line Versus Spot Ablation in Persistent Atrial Fibrillation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Prof. A. Schömig, Deutsches Herzzentrum Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. C00604
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): linear lesions to ablate persistent atrial fibrillation
  Interventions: Procedure: linear anatomically oriented ablations
- 2 (Experimental): focal electrophysiologically guided ablations to treat persistent atrial fibrillation
  Interventions: Procedure: focal electrophysiological oriented ablations

INTERVENTIONS:
Procedure: linear anatomically oriented ablations — linear lesions to ablate persistent atrial fibrillation
  Arms: 1
Procedure: focal electrophysiological oriented ablations — focal electrophysiologically guided ablations to treat persistent atrial fibrillation
  Arms: 2

SUMMARY:
In this randomized study dealing with the ablative treatment of persistent atrial fibrillation, two ablation strategies are compared: a more anatomically guided linear ablation scheme versus an electrophysiological guided focal ablation strategy aiming at the electrical isolating of the pulmonary veins and ablating areas of fragmented intracardiac electrograms thought to maintain atrial fibrillation.

DETAILED DESCRIPTION:
This randomized study deals with two different ablative treatment strategies for persistent atrial fibrillation: a more anatomically guided linear ablation scheme with encircling of the ipsilateral pulmonary veins (PV), a left atrial roof line and an anterior line bridging the anterior mitral anulus to the ostium of the left superior PV versus an electrophysiological guided focal ablation strategy aiming at isolating, electrically, the PV and ablating areas of fragmented intracardiac electrograms thought to maintain atrial fibrillation.

Both ablation approaches contain isolation of the most common source of triggering foci, i.e., the pulmonary veins and additional modification of the substrate maintaining atrial fibrillation.

The study endpoint is a combined efficacy/safety analysis. Extensive follow-up with three-monthly 7 days holter ECG is provided.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* symptomatic persistent (> 7 days lasting) atrial fibrillation
* at least one unsuccessful cardioversion or atrial fibrillation relapse in the first 3 months after cardioversion despite antiarrhythmic drug therapy
* oral anticoagulation (> 4 weeks prior to ablation)

Exclusion Criteria:

* moderate to severe valvular heart disease
* congenital heart disease
* LV-EF < 35%
* reversible cause for atrial fibrillation (e.g., hyperthyreosis)
* prior left atrial ablation or Maze operation
* left atrial thrombus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2004-08; Primary Completion 2008-05 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Sinus rhythm in follow-up | Sinus rhythm in follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Claus Schmitt, MD, Study Chair — Deutsches Herzzentrum Muenchen; Heidi Estner, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany